CLINICAL TRIAL: NCT06697457
Title: Comparison of the Effectiveness of Dynamic Isometric, Static Isometric and Craniocervical Flexor Exercise Training in Individuals with Chronic Neck Pain
Brief Title: Comparison of the Effectiveness of Different Exercise Types in Individuals with Chronic Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Ayşen Canan, Physiotherapist Ayşen Canan Pakeloğlu, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSKU-FTR-ACP-01
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-06

CONDITIONS: Chronic Neck Pain
Keywords: neck pain; chronic; exercise
MeSH Terms: conditions — Neck Pain; Bronchiolitis Obliterans Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: Four groups, parallel, randomized controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessors and patients were not informed about group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Conventional Treatment (Active Comparator): Conventional treatment will include electrotherapy agents (TENS, ultrasound and hotpack) and chin tuck posture exercises.
  Interventions: Other: Conventional Treatment Group
- Craniocervical Flexion Exercise Training (Active Comparator): Patients will receive exercise in addition to conventional treatment. The exercises will be performed with an air-filled pressure stabilizer placed in the sub-occipital region.
  Interventions: Other: Craniocervical Flexion Exercise Group; Other: Conventional Treatment Group
- Dynamic Isometric Exercise Training (Active Comparator): Patients will receive exercise in addition to conventional treatment. The exercises will be performed by the patient with an elastic band.
  Interventions: Other: Conventional Treatment Group; Other: Dynamic Isometric Exercise Group
- Static Isometric Exercise Training (Active Comparator): Patients will receive exercise in addition to conventional treatment. The patient will perform isometric exercises with maximal effort against neck flexion, extension, lateral flexion and rotation with his/her hand in a sitting position.
  Interventions: Other: Conventional Treatment Group; Other: Static Isometric Exercise Group

INTERVENTIONS:
Other: Craniocervical Flexion Exercise Group — The patient will first be taught to contract the deep cervical flexors. Patients will be placed in a supine position (without a pillow) to ensure a neutral neck position. Patients will be asked to perform slow, controlled head and upper cervical flexion by bringing the chin closer to the chest ("yes" movement). The stabilizer will be inflated to 20 mmHg. Gradual training will be given to increase the pressure value by 2 mmHg between 20 and 30 mmHg. Each pressure value (22, 24, 26, 28 mmHg) will be held for 10 seconds and repeated 10 times. The exercise will be performed with 10 repetitions, 10 seconds of contraction and 5 seconds of relaxation. Exercise training will begin with 20 mmHg and once the patient can hold it for 10 seconds with 10 repetitions, the next level on the pressure stabilizer will be moved on.Treatments will be performed 3 days a week for 8 weeks.
  Arms: Craniocervical Flexion Exercise Training
Other: Conventional Treatment Group — TENS will be applied with a TENS device at an intensity of 10-30 mA and a frequency of 80 Hz for 20 minutes. A pair of surface electrodes will be placed on the painful area of the neck. The intensity of TENS will be adjusted according to the patient's sensory thresholds so that the patient is not disturbed by a numb feeling. After TENS, continuous ultrasound will be applied to the cervical region to produce thermal effects. The intensity will be 1.5 W/cm² and the duration will be 5 minutes. Hotpack will be applied to the trapezius muscle for 10 minutes. Chin tuck exercise will be applied to the cervical region.Treatments will be performed 3 days a week for 8 weeks.
Other: Dynamic Isometric Exercise Group — The exercises will be performed by the patient with an elastic band. The progression of the exercises will be performed using different colors of Thera-bands with different resistances. It will start with the red Thera-band with the lowest resistance and then move on to the green and then blue Thera-bands with increasing resistance. Cervical isometric exercises will be performed with elastic resistance bands, maintaining the chin tuck position, forward, backward, crosswise, right and left. There will be 10 repetitions for 10 seconds for each. Progression in Therabands will be according to the patient. When the patient does 10 repetitions for 10 seconds, the next Theraband will be used.Treatments will be performed 3 days a week for 8 weeks.
  Arms: Dynamic Isometric Exercise Training
Other: Static Isometric Exercise Group — The patient will perform isometric exercises with maximal effort against neck flexion, extension, lateral flexion and rotation with his/her hand in a sitting position. Each exercise will be performed for 10 seconds, with 15-second breaks in between, for 10 repetitions. Each patient will start with submaximal resistance to help them adapt to isometric exercises, and then progress will be checked until the patient reaches the maximum resistance that can be tolerated by each session. It will consist of cervical flexion, cervical extension, right lateral flexion, left lateral flexion, right rotation, left rotation exercises. Progress in the exercises will be according to the Rating of Perceived Exertion Borg (RPE) Scale according to the weeks.Treatments will be performed 3 days a week for 8 weeks.
  Arms: Static Isometric Exercise Training

SUMMARY:
The aim of this study is to compare the effectiveness of craniocervical flexion, static and dynamic isometric exercise training applied with a conventional physiotherapy program in individuals with chronic neck pain.

DETAILED DESCRIPTION:
Neck pain is a significant musculoskeletal problem that is frequently encountered in society. Pain that cannot be diagnosed with a specific pathology is called "nonspecific" and pain that continues for more than three months is called "chronic pain". Chronic nonspecific neck pain has negative effects on function and quality of life. The importance of the exercise approach in the treatment of neck pain is quite great. Craniocervical flexion and static isometric exercises are frequently used in individuals with chronic neck pain. However, there are very few studies that include dynamic isometric exercises. The aim of this study is to compare the effectiveness of craniocervical flexion, static and dynamic isometric exercise training applied with a conventional physiotherapy program in individuals with chronic neck pain. The intervention groups of the study are deep cervical flexion exercise training, dynamic isometric exercise training and static isometric exercise training and electrotherapy group. The craniocervical flexion exercise training group will receive deep cervical flexor muscle training with Pressure Biofeedback, the dynamic isometric exercise group will receive exercise training with Thera-band, and the static isometric exercise group will receive neck isometric exercises. The electrotherapy group will receive hotpack, tens, and ultrasound applications. At the beginning and end of the study, pain, disability, posture, muscle strength, endurance, range of motion, and body awareness will be assessed in all individuals.TENS (Transcutaneous Electrical Nerve Stimulation) will be applied to all groups for 20 minutes with a TENS device at a strength of 10-30 mA and a frequency of 80 Hz. A pair of surface electrodes will be placed on the painful area of the neck. The intensity of TENS will be adjusted according to the patient's sensory thresholds so that they are not disturbed by a numbness sensation. After TENS, continuous ultrasound will be applied to the cervical region to produce thermal effects. The intensity will be 1.5 W/cm² and the duration will be 5 minutes. Hotpack will be applied to the trapezius muscle for 10 minutes. Chin tuck exercise will be applied to the cervical region.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 55,
* Scoring 15/50 or less on the Neck Disability Index,
* Having a history of chronic neck pain for at least 3 months,
* Having a pain level of 5/10 or more,
* Showing signs of cervical movement control dysfunction,
* Having cervical muscle tenderness during physical examination.

Exclusion Criteria:

* Being diagnosed with a vascular disease,
* Being diagnosed with a vestibular disease,
* Being diagnosed with hypertension,
* Being diagnosed with fibromyalgia or rheumatoid arthritis,
* Having had spine surgery in the last 12 months,
* Having received an exercise program or standard physiotherapy program involving the cervical region in the last 12 months,
* Having congenital or acquired kyphosis, scoliosis, etc. having postural deformity,
* Having specific neck pain such as cancer,
* Having fractures, instability, inflammatory diseases, history of neck trauma, infections, neurological deficit, having spinal diseases such as radiculopathy, spondylosis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Pain Assesment | 8 week
  The assessment will be made with Visual Analogue Scale (VAS) and algometer. VAS is considered both valid and reliable in measuring the pain intensity of patients. Each participant will be asked to indicate the intensity of pain they have experienced in the previous 24 hours. This will be done by marking on a 10 cm line where "0" is "No Pain" and "10" is "Maximum Pain".
Pain Assesment | 8 week
  An algometer with a 1 cm2 rounded surface area will be used for objective pain assessment. Measurements will be made on the spinous processes of C2 and c5 and the trapezius muscle. The assessor will gradually increase the pressure until pain or discomfort occurs and the patient says "yes". The average of the three measurements will be taken. A 30-second rest period will be given between each measurement.
Disability Assesment | 8 week
  Neck Disability Index, designed to assess how neck pain affects daily living activities, will be used. The questionnaire includes 10 items that measure disability secondary to neck pain. Scores range from 0-50 and are interpreted as follows:
  * 0-4 represents no disability,
  * 5-14 represents mild disability,
  * 15-24 represents moderate disability,
  * 25-33 represents severe disability,
  * 34 and above represents complete disability.

SECONDARY OUTCOMES:
Cervical Joint Range of Motion Assessment | 8 week
  Goniometer will be used for active ROM (flexion, extension, left/right rotation, left/right lateral flexion) measurements. Maximum ROM will be measured in degrees for each test. Participants will be asked to sit against the back of the chair, look forward, and position their arms in a relaxed manner.
Cervical Postur Assesment | 8 week
  Tragus Wall Distance Measurement will be performed with 2-3 practical trials to ensure that the participant has taken the correct posture. After the posture is appropriate, the tragus wall distance will be measured with a millimeter ruler while the participants stand naturally and perform cervical retraction
Cervical Postur Assesment | 8 week
  The craniovertebral angle will be measured for forward head posture in the sagittal plane. The craniovertebral angle will be measured with the photograph method. The camera is fixed 1.5 meters away on a flat surface aligned with the humeral head of the participants. The participants are asked to perform head flexion-extension movements to find the neutral head position and the participants are told to stay in the most appropriate position. A cursor is placed on the c7 spinous process and tragus in the photograph. The participants' photographs are taken 3 times. Craniovertebral angle is measured with the photographs taken and noted in degrees. The angles are averaged. Image processing will be done with Image J software
Cervical Strength Assessment | 8 week
  Hand Held dynamometer will be used for strength assessment. It will include 3 isometric contractions held for 3 seconds for flexion, extension, lateral flexion and rotation movements. The value greater than the maximal contractions will be recorded.
Cervical Endurance Assessment | 8 week
  In the Craniocervical Flexion Test, participants will be in a supine position and the compressed air unit will be placed behind the cervical spine, just below the occiput. It will be inflated to 20 mmHg initially and participants will be instructed to perform the craniocervical flexion movement. Thus, the pressure will increase to 22 mmHg and they will be asked to maintain this position for 10 seconds. Then, a 30-second rest period will be given and the entire procedure will be repeated for 24, 26, 28 and 30 mmHg. The final reading will be taken when the participant cannot hold the specific pressure for 10 seconds. Before the test, participants will be given enough time to practice.
Cervical Endurance Assesment | 8 week
  Cervical Flexion Endurance Test: Participants will be asked to lie in a crook-lying position. The physiotherapist will place their hand under the patient's head. They will be asked to lift their head approximately 2.5 cm off the bed and maintain this position for as long as possible. The test will end when the patient feels any pain or fatigue or when their head touches the therapist's hand. Endurance time was measured in seconds. The test will be performed twice with 3 minutes of rest between repetitions.
Cervical Endurance Assessment | 8 week
  Cervical Extensor Endurance Test: For the test, patients will be asked to lie in a prone position with their head and upper body positioned on the edge of the bed and their arms next to their body. A 2 kg sandbag will be placed on the patient's cervical region. They will then be asked to lift their head to a neutral position and maintain this position. The test will end when the patient feels any pain or fatigue or when there is a 5° deterioration in head position (measured with an inclinometer). The test will be repeated twice with a 3-minute rest interval and the longest holding time in seconds will be recorded as the test result.
Neck Awareness Assesment | 8 week
  It will be evaluated with the Fremantle Neck Awareness Questionnaire. It is a simple Likert-type questionnaire (0=Never/Never feel like this, 1= Rarely feel like this, 2= Sometimes or some of the time feel like this, 3= Often feel like this, 4= Always or most of the time feel like this) that evaluates the individual's altered perception. The questionnaire asks individuals 9 questions such as how they perceive their neck in relation to their body.

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Education and Research Hospital, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No